CLINICAL TRIAL: NCT03705442
Title: Probiotics as Adjuvant Therapy in the Treatment of Metastatic Colorectal Cancer: Randomized Double-blind Placebo-controlled Trial
Brief Title: Probiotics as Adjuvant Therapy in the Treatment of Metastatic Colorectal Cancer
Acronym: Probat-tmcc-17
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marin Golčić (Other)
Responsible Party: Sponsor-Investigator, Marin Golčić, Principal Investigator, University Hospital Rijeka
Organization: University Hospital Rijeka (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Probat-tmcc-17
Record Dates: First submitted 2018-02-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Loperamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: loperamide ("Seldiar")
- Probiotics (Experimental): Omni-Biotic 10
  Interventions: Dietary Supplement: Omni-Biotic 10; Drug: loperamide ("Seldiar")

INTERVENTIONS:
Dietary Supplement: Omni-Biotic 10 — All patients will have at their disposal current medications for diarrhea based on guidelines, and education regarding side effects and dietary recommendations will be undertaken. One cohort will also ingest a probiotic (OMNi-BiOTiC® 10AAD), while other cohort will take a placebo, same in colour, shape, taste and smell; both medications will be taken 2 per day, every 12 hours, over 84 days (6 chemotherapy cycles every 14 days).
  Other Names: OmniBiotic 10; Institut Allergosan
  Arms: Probiotics
Drug: loperamide ("Seldiar") — All the patients will have access to standard drugs for diarrhoea
  Other Names: loperamide ("Seldiar"), Standard antidiarrhoeal drug

SUMMARY:
The research will be prospective, randomised, placebo controlled and double-blinded.The research will be carried on with regards to Helsinki Declaration and following the guidelines of Good Clinical Practice.

DETAILED DESCRIPTION:
The investigators plan this research to be prospective, randomized, placebo-controlled and double blinded. It will be held according to Declaration of Helsinki and in harmony with Good Clinical Practice guidelines. All patients would be required to sign informed consent, approved by the Ethics Committee of Clinical Hospital Center (CHC) Rijeka.

All patients will have at their disposal current medications for diarrhea based on guidelines, and education regarding side effects and dietary recommendations will be undertaken. One cohort will also ingest a probiotic (OMNi-BiOTiC® 10AAD), while other cohort will take a placebo, same in colour, shape, taste and smell; both medications will be taken 2 per day, every 12 hours, over 84 days (6 chemotherapy cycles every 14 days). After 84 days, a regular examination will be undertaken. Total follow-up would be for two full cycles, at least 160 days. (Stool analyses will take place before and after chemotherapy(6-8 weeks after chemotherapy) and eventually three month later) Patients will be followed up in six main control points, t1, t2, t3, t4, t5, t6, which all represent the 1st day of matching 2-week-chemotherapy cycle. Each cycle starts exactly and at least 14 days from the first day of previous chemotherapy cycle. There would be no additional invasive procedures done for this study, regular blood examinations will be expanded with additional parameters. All patients would have the right to withdraw their written consent to participate in the study at any given time and for any reason whatsoever. (fecal analyses only before and 6-8 weeks after the last chemotherapy cycle)

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed diagnosis of colorectal cancer with metastasis;
* Patients older than 18 years of age;
* Patients starting first line of chemotherapy (FOLFIRI protocol);
* Signed patient consent form.

Exclusion Criteria:

* Present ileostomy;
* Decompensated patients;
* Terminal stage patients (<6 months life expectancy);
* Patients not mentally able to adhere to the protocol;
* Patients using >3 yoghurts per week or any other probiotics;
* Or any other condition which would not allow safe administration of the drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-02-09 (Estimated); Study Completion 2020-02-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade III/IV diarrhoea between the two groups of patients | 3 months
  To see whether application of OMNi-BiOTiC® 10 AAD probiotic will reduce grade III/IV diarrhea during the chemotherapy based on FOLFIRI protocol which would be followed by Bowel Movement Diary and Bristol Scale Stool Chart.

SECONDARY OUTCOMES:
Difference of zonulin concentration between the two groups of patients | 3 months
  To see whether the group on probiotics will have lower values of calprotectin and zonulin14
Difference of vitamin D concentration between the two groups of patients | 3 months
  To see whether the group on probiotics will have higher values of vitamin D (blood)
Difference in quality of life using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire core 30 (EORTC QLQ-C30) between the two groups of patients | 3 months
  To see whether the group on probiotics will have higher scores in EORCT QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Marin Golcic, MD, Principal Investigator — Clinical Hospital Center Rijeka
Locations (1):
- Department of Radiotherapy and Oncology, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided